CLINICAL TRIAL: NCT06271746
Title: A Prospective, Randomized, Double-blind, Sham-controlled Clinical Study Assessing the Safety and Efficacy of FibroNova for the Treatment of Fibromyalgia.
Brief Title: Treatment of Fibromyalgia With the FibroNova Neuromodulation Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCH101
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; Neuromodulation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment. Randomized, double-blind, sham-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment with active FibroNova device (Active Comparator): Treatment of Fibromyalgia pain and symptoms with active FibroNova device. Participants will treat with an active device twice a day.
  Interventions: Device: FibroNova (Active mode)
- Treatment with Sham FibroNova device (Placebo Comparator): Treatment of Fibromyalgia pain and symptoms with Sham FibroNova device. Participants will treat with a sham device twice a day.
  Interventions: Device: FibroNova (Sham mode)

INTERVENTIONS:
Device: FibroNova (Active mode) — FibroNova neurostimulator of conditional pain modulation (CPM)
  Arms: Treatment with active FibroNova device
Device: FibroNova (Sham mode) — FibroNova neurostimulator with an electrical output not intended for neurostimulation
  Arms: Treatment with Sham FibroNova device

SUMMARY:
Fibromyalgia (FM) is a chronic disorder that affects the musculoskeletal system, causing widespread pain, tenderness, and fatigue. It is estimated to affect 1-5% of the population. The primary symptom of fibromyalgia is widespread pain throughout the body, accompanied by tenderness and sensitivity to pressure.

Pharmacological treatments include drugs such as antidepressants, anticonvulsants, and painkillers. Another treatment option for fibromyalgia is the use of devices such as Quell. Other non-pharmacological treatment options for fibromyalgia include cognitive-behavioral therapy (CBT), biofeedback, and relaxation techniques.

Remote Electrical Neuromodulation (REN) is a non-pharmacological technology that induces subthreshold, non-painful neurostimulation signals that activate an endogenic pain-management system termed Conditioned Pain Modulation (CPM), to produce generalized pain relief in remote body areas. Multiple studies have shown that REN is safe and effective for the acute treatment of migraine in adults and adolescents, as well as migraine prevention.

The current study examines the safety and efficacy of REN technology, implemented via the FibroNova device for treating fibromyalgia pain and related symptoms.

DETAILED DESCRIPTION:
Background Fibromyalgia (FM) is a chronic disorder that affects the musculoskeletal system, causing widespread pain, tenderness, and fatigue. It is estimated to affect 1-5% of the population. The primary symptom of fibromyalgia is widespread pain throughout the body, accompanied by tenderness and sensitivity to pressure. Secondary symptoms include fatigue, sleep disturbances, cognitive difficulties, headaches, depression, and anxiety. The exact cause of fibromyalgia is unknown, but it is believed to involve a combination of neurobiological, genetic, and environmental factors.

There is no cure for fibromyalgia, and only a minority of fibromyalgia patients continue taking medications for more than a short period due to either lack of efficacy, side effects, or both. Pharmacological treatments include drugs such as antidepressants, anticonvulsants, and painkillers, and operate by modulating pain signals in the brain and nervous system. Another treatment option for fibromyalgia is the use of devices, such as the Quell device by Neurometrix 3. Other non-pharmacological treatment options for fibromyalgia include cognitive-behavioral therapy (CBT), biofeedback, and relaxation techniques 2.

Remote Electrical Neuromodulation (REN) is a non-pharmacological technology that induces subthreshold, non-painful neurostimulation signals that activate an endogenic pain-management system termed Conditioned Pain Modulation (CPM), to produce generalized pain relief in remote body areas. Multiple studies have shown that REN is safe and effective for the acute treatment of migraine in adults and adolescents, as well as migraine prevention.

The CPM system, which is deficient in patients with migraine, has been shown to be abnormal in fibromyalgia patients as well, suggesting that fibromyalgia patients could potentially benefit from activating the CPM via REN. The current study aims to examine the safety and efficacy of REN technology, implemented via the FibroNova device for the treatment of fibromyalgia pain and related symptoms.

The FibroNova device

The device is a wireless wearable battery-operated stimulation unit controlled by a smartphone software application. Treatments with FibroNova are self-administered by the user. The FibroNova device includes several main components:

* A pair of electrodes covered with hydrogel and a removeable protective film
* An electronic circuitry and a battery contained in a plastic case
* A software that includes firmware and a software application for mobile platforms
* An armband to improve the adhesiveness and enable a discreet treatment

The study design A prospective, randomized, double-blind, sham-controlled trial. The ratio between treatment and control groups will be 1:1, stratified by prior use of prescribed medications for FM (up to 2 vs. 3 or more). the following are considered as FM medications for the stratification: Dulloxetine, Pregabalin, Milnacipran, Amitriptyline.

The study will consist of two main phases and a voluntary open-label extension phase:

4-week baseline phase- in which participants will report their symptoms daily via an electronic app diary (with no intervention);

12-week intervention phase- in which eligible participants perform two treatments per day (using FibroNova/identical looking sham (placebo) device, according to randomization), and continue to report symptoms daily via the app.

12-week open-label extension phase (OLE)- upon completion of the intervention phase, eligible participants will be offered to participate in an additional voluntary 12-week period in which they will receive active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is 18-70.
2. Meets ACR 2010 Diagnostic Criteria for FM.
3. Naïve to Nerivio and to FibroNova devices.
4. Possesses the basic cognitive and motor skills needed to operate his/her own smartphone.
5. Must be able and willing to comply with the protocol.
6. Must be able and willing to provide written informed consent.

Exclusion Criteria:

1. Change in prescribed medications for pain and/or fibromyalgia in the two months prior to enrolment.
2. Pregnant or lactating.
3. Has other significant comorbidities or pain problem(s) or undergoing specific therapies that in the opinion of the investigator may confound the study assessments.(e.g. active inflammatory joint disease, including spondyloarthropathy, or active malignancy, excluding Basal cell carcinoma).
4. Newly diagnosed with fibromyalgia (under six months).
5. Is currently implanted with an electrical and/or neurostimulation device (e.g., cardiac pacemaker or defibrillator, vagus nerve neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator bladder stimulator or Occipital nerve stimulator).
6. Known uncontrolled epilepsy.
7. Active substance use disorder that could interfere with study participation.
8. Use of opioids during the 2 months prior to enrolment.
9. Has undergone nerve block (occipital or other) during the 2 months prior to enrolment.
10. Patients with severe depression, and/or suicidality
11. Is participating in any other clinical study.
12. Use of a neuromodulation device specifically indicated for FM ( e.g.Quell ) currently or in the 2 months prior to enrolment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean reduction in pain level during the last 14 days of the treatment phase (weeks 15 through 16) compare to the last 14 days of baseline phase (weeks 3 through 4) | 16 weeks
  Mean change, from the last two weeks (weeks 3-4) of the baseline phase to the last two weeks (weeks 15-16) of the intervention phase, in the 2-week average of daily self-reported pain severity scores on NRS (0 to 10) that is based on the FIQR pain item.
Device safety (rate of adverse events and device related adverse events) | 28 weeks
  The incidence of adverse events in general and by seriousness, severity and association to the device.

SECONDARY OUTCOMES:
Mean change in the Revised Fibromyalgia Impact Questionnaire FIQR total score | 16 weeks
  Mean change in the Revised Fibromyalgia Impact Questionnaire FIQR total score from the end of the baseline phase (end of week 4) to the end of the intervention.phase (end of week 16)
Mean change in FIQR functionality sub-scale score | 16 weeks
  Mean change in FIQR functionality sub-scale score from the end of the baseline phase (end of week 4) to the end of the intervention.phase (end of week 16)
Mean change in FIQR pain item score | 16 weeks
  Mean change in FIQR pain item score from the end of the baseline phase (end of week 4) to the end of the intervention.phase (end of week 16)
Mean change in Brief Pain Inventory (BPI) score | 16 weeks
  Mean change in Brief Pain Inventory (BPI) from the end of the baseline phase (end of week 4) to the end of the intervention.phase (end of week 16)
Improvement in patient global impression according to PGIC score | 16 weeks
  Percentage of participants who were categorized as "Improved (Very Much Improved, Much Improved, or Minimally Improved)" According to the Patient Global Impressions of Change (PGIC) at the end of week 12.
Mean reduction in functional disability during the last 14 days of the treatment phase (weeks 15 through 16) compare to the last 14 days of baseline phase (weeks 3 through 4) | 16 weeks
  Mean change, from the last two weeks of the baseline phase (weeks 3-4 to the last two weeks of the intervention phase (weeks 15-16), in the 2-week average of daily self-reported functional disability scores on NRS (0 to 10) that is based on the FIQR disability item.

OTHER OUTCOMES:
Improvement in quality of life | 16 weeks
  Mean change, from baseline to end of the intervention phase according to SF-36 quality of life questionnaire total score.
Improvement in sleep quality | 16 weeks
  Mean change, from the last two weeks of the baseline phase (weeks 3-4) to the last two weeks of the intervention phase (weeks 15-16), in the 2-week average of daily self-reported level of sleep quality, on an 11-level scale (based on the FIQR item), where 0 is "perfect sleep" and 10 is "could not sleep at all".
Mean change in level of depression | 16 weeks
  Mean change, from the last two weeks of the baseline phase (weeks 3-4) to the last two weeks of the intervention phase (weeks 15-16), in the 2-week average of daily self-reported level of depression on a 11-level scale (based on the FIQR item), where 0 is "not depressed at all" and 10 is "most depressed ever".
Mean change in level of anxiety | 16 weeks
  Mean change, from the last two weeks of the baseline phase (weeks 3-4) to the last two weeks of the intervention phase (weeks 15-16), in the 2-week average of daily self-reported level of anxiety, on a 11-level scale (based on the FIQR item), where 0 is "not anxious at all" and 10 is "most extremely anxious".
Mean change in level of cognitive impairment | 16 weeks
  Mean change, from the last two weeks of the baseline phase (weeks 3-4) to the last two weeks of the intervention phase (weeks 15-16), in the 2-week average of daily self-reported level of cognitive impairment on an 11-level scale (based on the FIQR item), where 0 is "no cognitive impairment at all" and 10 is "most severe impairment".
Mean change in level of cognitive presenteeism | 16 weeks
  Mean change, from the last two weeks of the baseline phase (weeks 3-4) the the last two weeks of the intervention phase (weeks 15-16), in the 2-week average daily self-reported occurrence of presenteeism on a dichotomous answer (based on the FIQR item), where 0 is "No, I felt as productive as usual at work (or school)" and 1 is "Yes, I felt greatly unproductive at work (or school).
Mean reduction of at least 30% in pain level | 16 weeks
  Percentage of patients with average reduction of 30% or more in pain intensity (NRS) - from the last two weeks of the baseline phase (weeks 3-4) the the last two weeks of the intervention phase (weeks 15-16).
Rate of treatment tolerability | 28 weeks
  Percentage of participants who indicated that the treatment was well tolerated or above, according to a multiple-choice question filled out at the end of the study (end of OLE/ upon withdrawal).
User experience | 28 weeks
  Percentage of participants that reported a positive user experience, based on the self-report user experience questions.
Patient Global Impression- change (PGI-C | 28 weeks
  Percentage of patients with an 'improved' PGI-C score at the end of week 12 of the intervention phase.
Patient Global Impression- change (PGI-C)- mid study: | 16 weeks
  Percentage of patients with an 'improved' PGI-C score at the mid-intervention phone call follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clauw, MD, Study Chair — University of Michigan
Locations (4):
- United States (3):
  - Clinical Research Professionals, Chesterfield, Missouri
  - ClinVest Headlands Research, Springfield, Missouri
  - Gershon Pain Specialists, Virginia Beach, Virginia
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No